CLINICAL TRIAL: NCT05034068
Title: Low Level Laser Therapy Versus Benzydamin in Prevention and Treatment of Oral Mucositis Induced by Anticancer Treatments (Clinical and Biochemical Study)
Brief Title: Low Level Laser Therapy Versus Benzydamin in Prevention and Treatment of Oral Mucositis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asem Mohammed Kamel Ali, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Treatment of Oral Mucositis
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Stomatitis (Oral Mucositis)
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): the patients will be treated by using oral care only and evaluation will be done before cancer treatment and weekly till the treatment completed. In each weekly visit, oral sites will be examined, and a score was given to each site based on the degree of mucositis.
- bezaydamine hydrochloride. (Active Comparator): All patients were advised to rinse 15 mL of the solution benzydamine for 2 min, four to eight times daily before and during, and for 2 weeks after completion of cancer therapy. In case of any problem (e.g. burning or stinging), patients will be allowed to dilute the solution with water in the ratio 1:1 or 1:2. Study evaluations will be conducted before cancer treatment and weekly thereafter until 2 weeks after completion of the therapy .In each weekly visit, oral sites were examined and a score was given to each site based on the degree of mucositis.
  Interventions: Drug: 0.15% bezaydamine hydrochloride.
- low-level laser therapy (Active Comparator): the patients will be treated by using a low-level laser therapy, the irradiations will be done three times a week using low power laser with a wavelength of 870 nm. The irradiation mode will be punctual and in contact, perpendicular to the oral mucosa. The power will be 60 mW, energy density of 6 J/cm2. Irradiation time will be 6 seconds per point based on the laser beam spot size of 0.55cm2. The irradiations will be done intra-orally avoiding the tumor site, oral examinations will be recorded at each irradiation session and the degree of mucositis will be recorded.
  Interventions: Device: low power laser with a wavelength of 870 nm

INTERVENTIONS:
Drug: 0.15% bezaydamine hydrochloride. — 0.15% bezaydamine hydrochloride was applied in oral mucosa in Patients with head and neck cancer under RT, CT treatment.
  Arms: bezaydamine hydrochloride.
Device: low power laser with a wavelength of 870 nm — the irradiations will be done three times a week using low power laser with a wavelength of 870 nm. The irradiation mode will be punctual and in contact, perpendicular to the oral mucosa. The power will be 60 mW, energy density of 6 J/cm2. Irradiation time will be 6 seconds per point based on the laser beam spot size of 0.55cm2
  Arms: low-level laser therapy

SUMMARY:
A prospective study will be conducted at the Department of Oral Medicine, Periodontology, Diagnosis and Oral Radiology Faculty of Dental Medicine, Assiut branch Al-Azhar University. Patients with head and neck cancer under RT, CT treatment participated in this study were selected from South Egypt Cancer Institute. During clinical examination the medical history of the patient will be recorded. Data related to base illness, type and stage of RT treatment, association or not to chemotherapy will be collected during the whole treatment. After clinical examination, the patients will receive a kit containing toothbrush, dentifrice, and subsequent oral hygiene instruction. Then the patients will be classified into 3 groups as follow: Group I (control group): the patients will be treated by using oral care only and evaluation will be done before cancer treatment and weekly till the treatment completed. Group II: the patients will be treated by using 0.15% bezaydamine hydrochloride. All patients were advised to rinse 15 mL of the solution benzydamine for 2 min, four to eight times daily before and during, and for 2 weeks after completion of cancer therapy. Group III: the patients will be treated by using a low-level laser therapy, the irradiations will be done three times a week using low power laser with a wavelength of 870 nm. The irradiation mode will be punctual and in contact, perpendicular to the oral mucosa.

ELIGIBILITY:
Inclusion Criteria:

-patients with head and neck carcinoma were scheduled to receive a RT treatment (two dimensional techniques), covering a wide area of the head and neck region, The RT protocol of the hospital for head and neck cancer patients consisted of treatment sessions 5 days a week, 2Gy per fraction, with a total dose of 70 Gy over 7 weeks (35 sessions). A minimum dose of 50 Gy was delivered to the oral cavity of all patients in the study, either exclusively or associated with chemotherapy.

Exclusion Criteria:

* Karnofsky performance status (KPS)less than 60% .
* Hypersensitivity to benzydamine or typical NSAIDs.
* Patients were excluded if they had lock jaw, any previous medical condition (s) hampering wound healing (e.g., diabetes mellitus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
TNF-α [picograms/millimeter (pg/ml)] in saliva | Change from Baseline (before Anti-cancer treatment) at 7 weeks (after Anti-cancer treatment)
  Unstimulated saliva (2 mL) were obtained after oral rinse with room-temperature water. It was be stored in sterile collection tubes that were labeled at - 80C. Enzyme-linked immunosorbent assays were used to quantify TNF-α amount in picograms.
IL-6 [picograms/millimeter (pg/ml)] in saliva | Change from Baseline (before Anti-cancer treatment) at 7 weeks (after Anti-cancer treatment)
  Unstimulated saliva (2 mL) were obtained after oral rinse with room-temperature water. It was be stored in sterile collection tubes that were labeled at - 80C. Enzyme-linked immunosorbent assays were used to quantify IL-6 amount in picograms.
WHO scale for severity of oral mucositis. | Change from Baseline (7 days after the beginning of Anti-cancer treatment) at 7 weeks (completion of Anti-cancer treatment)
  WHO scale scoring severity of oral mucositis by assessor as following:
  Score 0-no signs or symptoms. Score 1-oral soreness and erythema. Score 2-oral erythema and ulcers, both solid and liquid diets tolerated. Score3-oral ulcers, liquid diet only. Score 4-oral alimentation impossible.
National Institute of the Cancer-Common Toxicity criteria (NIC-CTC) RT-induced oral mucositis scale for extent of oral mucositis. | Change from Baseline (7 days after the beginning of Anti-cancer treatment) at 7 weeks (completion of Anti-cancer treatment)
  (NIC-CTC) RT-induced oral mucositis scale scoring extension of mucositid as following: (0) patients with oral mucosa presenting no visible alteration.
  1. Presence of erythema.
  2. Ulcers with up to 1.5 cm diameter and noncontiguous.
  3. Ulcers larger than 1.5 cm diameter and contiguous.
  4. Ulcers exhibiting necrosis and bleeding.
  5. Death related to toxicity
visual analog scale (VAS) scale for pain assessment | Change from Baseline (7 days after the beginning of Anti-cancer treatment) at 7 weeks (completion of Anti-cancer treatment)
  The VAS was modified according to the scale proposed by Bensadoun et al. : scores 1 and 2 (mild pain) were considered grade I, scores 3 and 4 (moderate pain) were grade II, scores of 5 to 7 (severe pain) were grade III and scores of 8 to 10 (very severe pain) were grade IV.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf I Gaafar, professor, Study Director — Faculty of dental medicine Al-Azhar university Assiut Branch; Azza sh Mahmoud, phD, Principal Investigator — South Egypt Cancer Institute, Assiut University.
Locations (1):
- Faculty of dental medicine Al-Azhar University (Assiut branch), Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sonis ST, Elting LS, Keefe D, Peterson DE, Schubert M, Hauer-Jensen M, Bekele BN, Raber-Durlacher J, Donnelly JP, Rubenstein EB; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Perspectives on cancer therapy-induced mucosal injury: pathogenesis, measurement, epidemiology, and consequences for patients. Cancer. 2004 May 1;100(9 Suppl):1995-2025. doi: 10.1002/cncr.20162. PMID 15108222
- [Background] Peterson DE. New strategies for management of oral mucositis in cancer patients. J Support Oncol. 2006 Feb;4(2 Suppl 1):9-13. PMID 16499139
- [Background] Guimaraes DM, Ota TMN, Da Silva DAC, Almeida FLDS, Schalch TD, Deana AM, Junior JMA, Fernandes KPS. Low-level laser or LED photobiomodulation on oral mucositis in pediatric patients under high doses of methotrexate: prospective, randomized, controlled trial. Support Care Cancer. 2021 Nov;29(11):6441-6447. doi: 10.1007/s00520-021-06206-9. Epub 2021 Apr 24. PMID 33893842